CLINICAL TRIAL: NCT00634881
Title: Consolidation Therapy With Alemtuzumab (MabCampath®) in Patients With Chronic Lymphocytic Leukemia Who Are in Complete or Partial 2nd Remission After Cytoreduction With Fludarabine or Fludarabine Plus Cyclophosphamide or Fludarabine Plus Cyclophosphamide Plus Rituximab or Bendamustine or Bendamustine Plus Rituximab - a Phase I/II Study
Brief Title: Alemtuzumab in Treating Patients With B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2i; CDR0000587746 (Other: Clinical Data Repository)
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: Alemtuzumab i.v. (Experimental): Intravenous administration of alemtuzumab according to the 3 + 3 dose escalation design.
  Interventions: Biological: Alemtuzumab i.v.
- Cohort B: Alemtuzumab s.c. (Experimental): After i.v. MTD (maximum tolerable dosage) has been determined, subcutaneous dose escalation is performed according to the same escalation rules as for cohort A, starting with the recommended dose level of i.v. application.
  Interventions: Biological: Alemtuzumab s.c.

INTERVENTIONS:
Biological: Alemtuzumab i.v. — Alemtuzumab will be administered once per week as a 2 h infusion
  * Dose level I: 10mg once weekly (start with dose escalation : 3 mg on day 1, 10mg on day 2) Duration
  * Dose level II: 20mg once weekly (start with dose escalation: 3mg on day 1, 10mg on day 2, 20mg on day 3)
  * Dose level III: 30mg once weekly (start with dose escalation: 3mg on day 1, 10mg on day 2, 30mg on day 3)
  Arms: Cohort A: Alemtuzumab i.v.
Biological: Alemtuzumab s.c. — Alemtuzumab will be administered once per week subcutaneously
  * Dose level I: 10mg once weekly (start with dose escalation : 3 mg on day 1, 10mg on day 2) Duration
  * Dose level II: 20mg once weekly (start with dose escalation: 3mg on day 1, 10mg on day 2, 20mg on day 3)
  * Dose level III: 30mg once weekly (start with dose escalation: 3mg on day 1, 10mg on day 2, 30mg on day 3)
  Arms: Cohort B: Alemtuzumab s.c.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This phase I/II trial is studying the side effects and best dose of alemtuzumab in treating patients with B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the safest dose of alemtuzumab as consolidation therapy in patients in second remission after fludarabine phosphate alone; fludarabine phosphate and cyclophosphamide; fludarabine phosphate, cyclophosphamide, and rituximab; bendamustine hydrochloride alone; or bendamustine hydrochloride and rituximab.
* To determine the frequency of cytomegalovirus reactivations or infections during or after alemtuzumab treatment.
* To determine which dose of alemtuzumab is efficient to eliminate minimal residual disease in peripheral blood and bone marrow (i.e., to turn a clinical partial remission into a clinical complete remission [CR], to turn a flow cytometry-positive CR into a flow cytometry-negative CR, or to turn a PCR-positive CR into a PCR-negative CR).
* To determine the pharmacokinetic profile of alemtuzumab.
* To compare the pharmacokinetic profile between intravenous versus subcutaneous administration of alemtuzumab.

OUTLINE: This is a multicenter, dose-escalation study of alemtuzumab.

* Group 1: Patients receive escalating doses of alemtuzumab IV over 2 hours once weekly for 8 weeks until the maximum tolerated dose (MTD) is determined.
* Group 2: Patients receive escalating doses of alemtuzumab subcutaneously once weekly for 8 weeks, beginning with the MTD determined in group 1 until a second MTD is determined.

Patients undergo bone marrow and blood sample collection periodically for laboratory and pharmacokinetic studies. Samples are analyzed for minimal residual disease and T-cell subsets (i.e., CD4 and CD8) via quantitative-PCR analysis and flow cytometry and cytomegalovirus antigens via PCR.

After completion of study treatment, patients are followed at 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of B-cell chronic lymphocytic leukemia (B-CLL)
* Disease in complete or partial remission after completion of 4-6 courses of second-line cytoreductive therapy no less than 90 days and no more than 150 days ago

  * Second-line cytoreductive therapy must comprise 1 of the following regimens:

    * Fludarabine phosphate alone (F)
    * Fludarabine phosphate and cyclophosphamide (FC)
    * Fludarabine phosphate, cyclophosphamide, and rituximab (FCR)
    * Bendamustine hydrochloride alone (B)
    * Bendamustine hydrochloride and rituximab chemotherapy (BR)
* Complete minimal residual disease response defined by the following:

  * At least negativity of 4-color-cytometry and/or even PCR-amplifiable clonal CDR III rearrangement of the IgV_H

    * For PCR analysis, blood sample need to be taken at beginning or during second-line cytoreductive therapy before achievement of a clinical complete remission
* Disease not refractory to first-line F/FC/FCR/B/BR if received such therapy

Exclusion criteria:

* Presence of bulky lymph nodes (> 5 cm) after second-line F/FC/FCR/B/BR
* Clinically apparent autoimmune cytopenia (i.e., autoimmune hemolytic anemia, autoimmune thrombocytopenia, or pure red cell aplasia)
* CNS involvement with B-CLL

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* ANC ≥ 1,500/µL
* Platelets ≥ 50,000/µL
* Creatinine ≤ 1.5 times the upper normal limit (ULN)
* Conjugated bilirubin ≤ 2 times ULN
* Thyroid function normal
* Not pregnant or nursing
* Fertile patients must use effective contraception

Exclusion criteria:

* Severe infection during second-line treatment with F/FC/FCR/B/BR, meeting any 1 of the following criteria:

  * Any episode of NCI grade 4 infection
  * More than 1 episode of NCI grade 3 infection
* Medical condition requiring long-term use of oral corticosteroids for more than 1 month
* Active bacterial, viral, or fungal infection
* HIV, hepatitis B virus, and/or hepatitis C virus-positive serum status
* Concurrent severe diseases that exclude the administration of protocol therapy, including any of the following:

  * NYHA class III-IV heart insufficiency
  * Severe chronic obstructive lung disease with hypoxemia
  * Severe ischemic cardiac disease
* Active secondary malignancy other than B-CLL prior to the study
* Known hypersensitivity or anaphylactic reaction against murine proteins or one of the drug components

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 2 prior chemotherapies, including F/FC/FCR/B/BR therapy
* No more than 1 pretreatment (before second-line therapy) with chlorambucil or F/FC/FCR/B/BR
* No chemotherapy or radiotherapy for any neoplastic disease other than B-CLL prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-11; Primary Completion 2010-01 (Actual); Study Completion 2012-02-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 28 days after the last dose of study medication
  • Dose-limiting toxicity (DLT) and maximal tolerable dose (MTD) DLT is defined as a) all grade III/IV non-hematologic toxicity and b) all grade IV hematologic toxicity lasting for more than 2 weeks (excluding lymphopenia) occuring during or within 4 weeks after end of consolidation therapy.
Maximum tolerated dose | 28 days after the last dose of study medication
  • Dose-limiting toxicity (DLT) and maximal tolerable dose (MTD) DLT is defined as a) all grade III/IV non-hematologic toxicity and b) all grade IV hematologic toxicity lasting for more than 2 weeks (excluding lymphopenia) occuring during or within 4 weeks after end of consolidation therapy.

SECONDARY OUTCOMES:
Rate of complete minimal residual disease response | will be tested repeatedly, first time 3 months after the last dose of study medication, last time point 24 months after last dose of study medication
  • Rate of molecular responses (defined by negativity of 4- colour- cytometry in BOTH peripheral blood AND bone marrow in patients in clinical CR) The approved laboratory diagnostics for detection of MRD response is 4-colour flow cytometry. Collaterally, it is possible to take samples for potential PCR- analysis for confirmation if available.
Rate of immunophenotypic remission using 4-color flow cytometry | will be tested repeatedly, first time 3 months after the last dose of study medication,
Rate of infections (especially CMV infections and reactivations) | upt to 24 months after last dose of study medication (end of study)
Rate of severe hematologic and non-hematologic side effects | 28 days after the last dose of study medication
Pharmacokinetics of alemtuzumab (after IV and subcutaneous administration) | up to 8 weeks during the alemtuzumab treatment
  Pharmacokinetic samples will be taken at week 4 and 8 during alemtuzumab treatment at the following time points: 0, 4, 8, 24, 48, 96, 168 h
Progression-free survival | upt to 24 months after last dose of study medication (end of study)
Overall survival | upt to 24 months after last dose of study medication (end of study)
Complete remission rate | 28 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (6):
- Germany (6):
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Klinikum Barnim GmbH, Werner Forssmann Krankenhaus, Eberswalde
  - Universitatsklinikum Heidelberg, Heidelberg
  - Klinikum Lippe - Lemgo, Lemgo
  - III Medizinische Klinik Mannheim, Mannheim
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Sawaf O, Fischer K, Herling CD, Ritgen M, Bottcher S, Bahlo J, Elter T, Stilgenbauer S, Eichhorst BF, Busch R, Elberskirch U, Abenhardt W, Kneba M, Hallek M, Wendtner CM. Alemtuzumab consolidation in chronic lymphocytic leukaemia: a phase I/II multicentre trial. Eur J Haematol. 2017 Mar;98(3):254-262. doi: 10.1111/ejh.12825. Epub 2016 Dec 1. PMID 27862308